CLINICAL TRIAL: NCT01922960
Title: Microcirculatory Assessment in Patients With Trauma and Severe Burns
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: investigators decided not to move forward with project
Sponsor: University of South Alabama (Other)
Responsible Party: Principal Investigator, William Richards, Study Chair and Principle Investigator, University of South Alabama
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: 12-092
Record Dates: First submitted 2013-06-27; First posted 2013-08-14 (Estimated); Last update posted 2017-11-29 (Actual); Status verified 2017-11

CONDITIONS: Burns; Trauma
Keywords: trauma; multiple organ dysfunction syndrome
MeSH Terms: conditions — Burns; Wounds and Injuries; Multiple Organ Failure

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- micro-imaging (Other): Sublingual or subconjunctival micro-imaging of the microcirculation taken for 3 minute intervals at certain timepoints.
  Timepoints for burn/trauma subjects: Day0, Day1,Day2,Day6 & Day7 Timepoints for general surgery population: post-induction, prior to resection, after resection,& closing of surgical wound.
  Interventions: Other: micro-imaging

INTERVENTIONS:
Other: micro-imaging — micro-imaging

SUMMARY:
Predict the development of multiple organ failure in patients with trauma and severe burns.

DETAILED DESCRIPTION:
Microvascular alterations are frequently seen in patients with sepsis, trauma, burns and those who are hemodynamically uncompensated(Shock).

The use of the Microscan is a non-invasive approach to visualize and assess impaired mucosal microcirculation in order to identify early on patients who are predisposed for MOF (multiple organ failure)

ELIGIBILITY:
Inclusion Criteria:

* Patients with severe burns/trauma ages 19-80. Patients undergoing elective abdominal or cardiothoracic surgery ages 19-69 years old

Exclusion Criteria:

* Patients undergoing elective surgery < 19 years old.

Ages: 19 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2012-04-07 (Estimated); Primary Completion 2014-02 (Actual); Study Completion 2014-02 (Actual)

PRIMARY OUTCOMES:
dysfunctional capillary density correlates with development of multiple organ failure | approximately 1 year to assess outcome measure

CONTACTS AND LOCATIONS:
Overall Officials: William O Richards, MD, Study Chair — University of South Alabama, Department of Surgery
Locations (1):
- University of South Alabama Medical Center, Mobile, Alabama, United States